CLINICAL TRIAL: NCT03089892
Title: A Perspective Study of Cancer-related Fatigue in Gynecologic Cancer Patients Under Chemotherapy
Status: Completed | Type: Observational
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Cheng-Chang Chang, Chief of Division, China Medical University Hospital
Other Study IDs: CRF-TSGH02
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Gynecologic Cancer; Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gynecologic cancer patients: Gynecologic cancer patients under chemotherapy

SUMMARY:
Chemotherapy is effective and most often used to treat cancer. The common drugs used on gynecologic cancer treatment include platinum compounds like cisplatin and carboplatin, which combined with taxane, topotecan, or liposomal doxorubicin to date. The most side effects of chemotherapy are esophagitis, mucositis, anxiety, nausea, vomiting, abdominal convulsion, painful swallowing, fatigue and sometimes diarrhea, dizziness, allergy (rash, itching), neutropenia, thrombocytopenia (fever, chills, cough, pain), anemia and bleeding.

Cancer-related fatigue (CRF), an indicator of quality of life, is a highly prevalent symptom (75-80%) during treatment and in patients with advanced cancer, yet is sometimes ignored. Fatigue affected their life more than pain. Proposed criteria for CRF have been adopted for inclusion in the International Statistical Classification of Disease and Related Health Problems, Tenth Revision, Clinical Modification (ICD-10-CM). Therefore, more in-depth researches on CRF are needed in Taiwan. Patients with CRF in need of improvement, commonly use nutrition supplements, acupuncture, healthy food, massage, drugs, etc. Hence, patients with CRF could consult their vital physician for an appropriate treatment. Furthermore, several drugs could be chosen to relieve CRF, including anemia drugs, antipsychotics or Astragalus polysaccharides extract.

The objective of this retrospective study is to collect and analyze the medical records of gynecologic cancer patients who who had received chemotherapy with or without prescription drug treatment for cancer-related fatigue in the Department of Obstetrics & Gynecology of Tri-Service General Hospital. This study will compare the fatigue improvement profile by different chemotherapy regimens, tumor stage, CRF treatment, etc. and investigate the association between the profile of fatigue improvement and fatigue cluster (weight loss and other symptoms of functional assessment of cancer therapy). This study will also collect blood specimens and analyze the correlation of the cytokine profile and/or immune profile.These results will supply physicians with more understanding about CRF, and help them to enhance the quality on gynecologic cancer care to being perfected in the future.

DETAILED DESCRIPTION:
About 60 gynecologic cancer patients' medical records are expected to collect and analyze in this retrospective study. The data collection from medical records of gynecologic cancer patients who had received chemotherapy with or without prescription drug treatment for cancer-related fatigue include the demographic information (e.g., height, weight, age, sex, tumor stage, time from tumor diagnoses, prescription drug of cancer-related fatigue treatment and chemotherapy toxicities), the diagnosis and severity of cancer-related fatigue, functional assessment of cancer therapy and so on.

ELIGIBILITY:
Inclusion Criteria:

* Gynecologic cancer patients under chemotherapy.
* aged 20 and above.

Exclusion Criteria:

* Patients who had been enrolled for other investigational drug trials within the data collection period of this study.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynecologic cancer
Study Population: Gynecologic cancer patients had accepted prescription drug treatment for cancer-related fatigue under chemotherapy in the Department of Obstetrics & Gynecology of Tri-Service General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Cancer-related fatigue evaluation by brief fatigue inventory-Taiwanese form(BFI-T) | Change from baseline cancer-related fatigue at each chemotherapy cycle (each cycle is 21 or 28 days)
  BFI was commonly used to evaluate the cancer-related fatigue during the clinical practice.

SECONDARY OUTCOMES:
Quality of life assessments by functional assessment of cancer therapy-general 7 (FACT-G7) | Change from baseline Quality of life at each chemotherapy cycle (each cycle is 21 or 28 days)
  FACT-G7 was usually used to assess the quality of life of cancer patients during the clinical practice.

OTHER OUTCOMES:
Cytokine and immune markers | Change from baseline cytokine and immune index at each chemotherapy cycle (each cycle is 21 or 28 days)
  Cytokine and immune markers will be assessed from blood of cancer patients during the each chemotherapy cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Chang Chang, M.D., Ph.D., Principal Investigator — China Medical University Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No